CLINICAL TRIAL: NCT01860820
Title: The Effect of Neuromuscular Stimulation on Post-Transplant Leg Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103618
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Kidney Transplant; Kidney Pancreas Transplant; Edema
Keywords: IPC/TEDS; Geko device
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best Medical Therapy (No Intervention): Participants will follow standard post-transplant protocols with IPC
- Geko device (Active Comparator): Participants will be fitted with the device to ensure that it functions according to the manufacturer's instructions by a trained technician. This device will be changed every 24 hours. The device is worn on both legs and is worn for 24 hours a day. The device will first be put on the first day following the day of surgery and will then be changed the following day at the same time for a total of 7 days after surgery.
  Interventions: Device: Geko device

INTERVENTIONS:
Device: Geko device
  Arms: Geko device

SUMMARY:
This will be a randomized, controlled trial involving kidney and kidney pancreas transplant patients. There will be 2 groups and patients that will be randomized to one of the two groups. Clinical outcomes will be compared for those in each group and clinical differences between patients who receive routine medical therapy with IPC/TEDS versus the Geko device will also be evaluated.

DETAILED DESCRIPTION:
This will be a randomized, controlled trial involving kidney and kidney pancreas transplant patients. There will be 2 groups and patients will be randomized to one of the two; one will receive standard of care IPC or TED stockings to help with circulation, the other group will use the geko device which is a newer device with Health Canada approval. Clinical outcomes will be compared for those in each group and clinical differences between patients who receive routine medical therapy with IPC/TEDS versus the Geko device will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 18 years old
* Undergoing kidney or kidney pancreas transplant surgery as the recipient
* Able and willing to provide written informed consent
* Absence of known peripheral vascular disease
* Body Mass Index of between 18 and 34
* Leg circumference at site of geko™ device placement is 24" or less

Exclusion Criteria:

* History of deep vein thrombosis
* Temporary or permanent cardiac pacing
* Patient is pregnant
* Any patient which may be excluded by way of warnings in the Manufacturer's Instructions for Use
* Any patient who requires an ECG electrode applied on the leg for continuous monitoring throughout therapy
* Previous leg(s) amputation
* Presence of any of the following in the site of intended device placement: cancerous lesion, swollen or infected or inflamed areas or skin eruptions i.e. phlebitis, thrombophlebitis, varicose veins
* History or signs of haematological disorders (especially in relation to clotting or coagulation disorders) including presence or history of thrombus formation
* BMI index >36
* Patients with any neurological disorder or disease that would interfere with proper assessment and or conduct of the trial
* History of implantable brain or other stimulator
* Patients who can not tolerate the stimulation from the GEKO device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Decrease in edema | Within 30 days post-transplant
  As measured by patient weight and leg diameter

SECONDARY OUTCOMES:
Patient satisfaction | 3 and 6 days after transplant
  Patients will be asked to complete a questionnaire at these time points to assess their satisfaction

OTHER OUTCOMES:
Use of diuretics | Within 30 days of transplant
  Diuretic use wil be tracked for participants in each of the arms to assess wither there is a difference.

CONTACTS AND LOCATIONS:
Overall Officials: Alp Sener, MD, Principal Investigator — Lawson Health Research Institute, London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No